CLINICAL TRIAL: NCT04525599
Title: A Phase 1, Randomized, Single Dose, Blinded, Dose-Escalation Study to Assess Safety, Tolerability and Immunogenicity of ASP3772, a Pneumococcal Vaccine, in Toddlers 12 to 15 Months of Age in Comparison to an Active Comparator
Brief Title: A Study to Assess the Safety, Tolerability and Immunogenicity of ASP3772, a Pneumococcal Vaccine, in Toddlers 12 to 15 Months of Age in Comparison to an Active Comparator
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affinivax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 3772-CL-2001; 2019-004503-12 (EudraCT Number)
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers; Pneumococcal Disease
Keywords: Pneumococcal Disease; ASP3772; Pneumococcal vaccine; Vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1, ASP3772 Low Dose (Experimental): Participants will receive a single intramuscular injection of ASP3772 administered on Day 1 at a low-dose level.
  Interventions: Biological: ASP3772
- Group 1, PCV13 Comparator (Active Comparator): Participants will receive a single intramuscular injection of the approved dose of PCV13 on Day 1.
  Interventions: Biological: PCV13
- Group 2, ASP3772 Medium Dose (Experimental): Participants will receive a single intramuscular injection of ASP3772 administered on Day 1 at a medium-dose level.
  Interventions: Biological: ASP3772
- Group 2, PCV13 Comparator (Active Comparator): Participants will receive a single intramuscular injection of the approved dose of PCV13 on Day 1.
  Interventions: Biological: PCV13
- Group 3, ASP3772 High Dose (Experimental): Participants will receive a single intramuscular injection of ASP3772 administered on Day 1 at a high-dose level.
  Interventions: Biological: ASP3772
- Group 3, PCV13 Comparator (Active Comparator): Participants will receive a single intramuscular injection of the approved dose of PCV13 on Day 1.
  Interventions: Biological: PCV13

INTERVENTIONS:
Biological: ASP3772 — Intramuscular (IM) injection
  Arms: Group 1, ASP3772 Low Dose; Group 2, ASP3772 Medium Dose; Group 3, ASP3772 High Dose
Biological: PCV13 — Intramuscular injection
  Other Names: Prevnar 13
  Arms: Group 1, PCV13 Comparator; Group 2, PCV13 Comparator; Group 3, PCV13 Comparator

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of three dose levels of ASP3772 in comparison to the active comparator Prevnar 13® (PCV13) in toddlers who have previously been administered the routine three-dose series of PCV13.

This study will also evaluate the immunogenicity (production of an immune response) of three different dose levels of ASP3772 in comparison to the active comparator PCV13 in toddlers who have previously been administered the routine three-dose series of PCV13.

DETAILED DESCRIPTION:
After screening, participants will be randomized to ASP3772 or PCV13 on Day 1. A single dose of ASP3772 will be administered on Day 1 as an injection into the right or left thigh muscle at one of three dose levels. The participants randomized to PCV13 will receive a single intramuscular injection of the approved dose of PCV13 into the right or left thigh muscle. All participants will remain at the study site for approximately 30 to 60 minutes following vaccination in order for study site personnel to evaluate any immediate reactions, if needed. The participant's parent/legal guardian will observe for reactions, including daily body temperature measurements and tolerability assessments, from Day 2 through Day 7 and record observed events in the electronic diary device.

All participants will have study visits on Day 7 (+ 1 day) and Day 30 (± 5 days) post-vaccination. The Day 7 visit may be conducted on site or by telephone call.The end-of-study visit will occur on Day 180 (± 14 days), which will be a safety follow-up by telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy toddler who has previously completed a 3-dose infant series of PCV13 with the last vaccination greater than 2 months prior to study vaccination.
* Subject is afebrile within the last 48 hours (temperature measured orally is < 100 °F [37.8°C]; measured rectally or tympanic is < 101 °F [38.3°C]; measured in an axillary position or temporal is < 98.4 °F [36.9°C]).
* Subject's parent/legal guardian is able to read, understand and complete study questionnaires (i.e., the electronic subject diary device).
* Subject's parent/legal guardian along with the subject is able and is willing to attend all scheduled visits and to comply with the study procedures.
* Subject's parent/legal guardian has access to a telephone.
* Subject's parent/legal guardian agrees not to enroll subject in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has a known hypersensitivity to any vaccine.
* Subject has an immune disorder(s) (including autoimmune disease) and/or clinical conditions requiring immunosuppressive drugs, known or suspected impairment of immunological function or a history of congenital or acquired immunodeficiency.
* Subject has or his/her mother has known human immunodeficiency virus infection or known to be hepatitis B surface antigen-positive.
* Subject has functional or anatomic asplenia.
* Subject has known neurological or cognitive behavioral disorders including clinically significant developmental disorder and related disorders.
* Subject has any evidence of any unstable or active clinically significant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease.
* Subject has any active malignancy or history of malignancy.
* Subject has been in receipt of intramuscular, oral, intravenous, inhaled or intranasal corticosteroid treatment within 2 weeks prior to study vaccination or is planned to receive these medications within 4 weeks after study vaccination. Note: Use of topical corticosteroids is permitted.
* Subject has received any live-attenuated vaccines within 4 weeks prior to receipt of the study vaccine or inactivated vaccines within 2 weeks prior to receipt of study vaccine.
* Subject has previously received an approved (other than PCV13) or investigational pneumococcal vaccine.
* Subject has had any prior receipt of a blood transfusion or blood products, including immunoglobulins.
* Subject has received investigational therapy within 30 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has received a systemically absorbed antibacterial agent within 7 days prior to study vaccination.
* Subject has a history of microbiologically-proven invasive disease caused by S. pneumoniae.
* Subject has received acetaminophen or nonsteroidal anti-inflammatorydrugs (NSAIDs) within 24 hours prior to receipt of study vaccine.
* Subject has a coagulation disorder.
* Subject's parent/legal guardian is unlikely to adhere to study procedures, keep appointments, or is planning to relocate during the study and the subject cannot be adequately followed for safety according to the protocol.
* Subject who has a condition which makes the subject unsuitable for study participation.
* Subject's parent(s)/legal guardian is an employee of Astellas Pharma Global Development Inc., the study-related contract research organizations (CROs), or the study site.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to Day 30
  A TEAE is defined as an adverse event (AE) observed after study vaccination and up to 30 days post-vaccination. A vaccine-related TEAE is defined as any TEAE with a causal relationship assessed as "yes" by the investigator.
Number of Participants With Body Temperature Abnormalities and/or Adverse Events | Up to Day 30
  Number of participants with potentially clinically significant body temperature abnormalities.
Reactogenicity Assessed by Number of Solicited Local Reactions | Up to Day 7
  Local reactions are tenderness, movement restriction, redness/erythema and swelling and induration. Local reactogenicity will be evaluated at approximately 30 to 60 minutes post-dose by study site personnel and recorded in an electronic diary device by the participant's parent/legal guardian while at the study site on day 1. The participant's parent/legal guardian will observe reactogenicity and tolerability from day 2 through day 7, and record observed events daily in the electronic diary device. Grades range from 1 (mild) to 4 (potentially life-threatening).
Reactogenicity assessed by Number of Solicited Systemic Reactions | Up to Day 7
  Systemic reactions are vomiting, diarrhea, fever, irritability, decrease of appetite and increase or decrease in sleep. Body temperature will be assessed pre-dose and approximately 30 to 60 minutes post-dose. The participant's parent/legal guardian will be asked to observe the systemic reactogenicity symptoms from day 2 through day 7 and record observed events daily in the electronic diary device. Grades range from 1 (mild) to 4 (potentially life-threatening).

SECONDARY OUTCOMES:
Proportion of Participants Achieving a Serotype-specific Anticapsular Polysaccharide Immunoglobulin G (PS IgG) Concentration of ≥ 0.35 µg/mL for ASP3772 | Up to 30 days
  PS IgG concentration measure will be used to characterize the immunological response 30 days following administration of ASP3772.
Proportion of Participants Achieving a Serotype-specific Anticapsular PS IgG Concentration of ≥ 0.35 µg/mL for PCV13 | Up to 30 days
  PS IgG concentration measure will be used to characterize the immunological response 30 days following administration of PCV13.
Proportion of Participants Achieving a Serotype-specific Opsonophagocytic Activity (OPA) Antibody Titer ≥ 1:8 for ASP3772 | Up to 30 days
  OPA measure will be used to characterize the immunological response 30 days following administration of ASP3772.
Proportion of Participants Achieving a Serotype-specific OPA Antibody Titer ≥ 1:8 for PCV13 | Up to 30 days
  OPA measure will be used to characterize the immunological response 30 days following administration of PCV13.
Geometric Mean Titer (GMT) for Serotype-specific OPA for ASP3772 | Up to 30 days
  OPA measure will be used to characterize the immunological response 30 days following administration of ASP3772.
Geometric Mean Titer (GMT) for Serotype-specific OPA for PCV13 | Up to 30 days
  OPA measure will be used to characterize the immunological response 30 days following administration of PCV13.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (17):
- United States (17):
  - Dermatology Trial Associates, Bryant, Arkansas
  - The Childrens Clinic, Jonesboro, Arkansas
  - Emmaus Research Center, Inc, Anaheim, California
  - Madera Family Medical Group, Madera, California
  - Ctr Clin Trials San Gabriel, West Covina, California
  - Gentle Medicine Associates, Boynton Beach, Florida
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - PMG Research, Statesville, North Carolina
  - Oklahoma State University Center for Health Sciences, Tulsa, Oklahoma
  - Pediatrics Medical Associates, East Norriton, Pennsylvania
  - Coastal Pediatric Associates, Charleston, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Clinical Research Associates, Houston, Texas
  - Tanner Clinic, Layton, Utah
  - Pediatric Care, Provo, Utah
  - MultiCare Institute, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial as it meets one or more of the exceptions described on www.clinicalstudydatarequest.com under "Sponsor Specific Details for Astellas."